CLINICAL TRIAL: NCT05081778
Title: Dissociative Disorders in Obesity
Brief Title: Dissociative Disorders in Obesity (Dissobe)
Acronym: Dissobe
Status: Completed | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02797-48
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Dissociative Disorder
MeSH Terms: conditions — Obesity; Dissociative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patient following a medical course
  Interventions: Behavioral: Obese patient following a medical course
- Obese patient following a surgical course
  Interventions: Behavioral: Obese patient following a medical course

INTERVENTIONS:
Behavioral: Obese patient following a medical course — Questionnaires for the assessment of dissociative disorders in obese patients : DES scale of Carlson and Putman, SDQ-20 of Nijenhuis, comorbidities, Dutch Eating Behaviour Questionnaire (DEBQ), questionnaire of Rosenberg

SUMMARY:
THe aim of this study is to determine the frequency of dissociative tendencies in the obese population treated at the CELIOBE (Liberal Center for Obesity Support) at Hôpital Privé La Louvière among patients consulting for the first time and looking for a medical or surgical course. The DES scale of Carlson and Putman will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Obesity defined by a Body Mass Index (BMI) ≥ 30 kg / m2
* Patient seen in consultation at CELIOBE for the first time for the management of an overweight problem, wishing for surgical or medical care
* Patient having been informed and not opposing to this research
* Patient affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Psychotic antecedents: Schizophrenia, Schizoaffective disorders, Hallucinatory psychoses, Brief psychotic attacks
* Addictive behaviors (alcohol, drug addiction)
* Drug use
* Taking antipsychotics and mood stabilizers
* Dissociative identity disorders proven
* Bipolar disorders or severe mental illness
* Understanding troubles
* Protected patient: Major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision; Hospitalized without consent
* Pregnant, breastfeeding or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese population with a body mass index over 30kg/m2 Minimum age : 18 years-old Patients consulting for the first time at CELIOBE and wishing a medical or surgical course.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
The degree of dissociative tendencies | 1 day
  The degree of dissociative tendencies measured by the Carlson and Putman DES scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé La Louvière, Lille, Haut de France, France